CLINICAL TRIAL: NCT06786585
Title: Extended Clinical Follow up and Biospecimen Collection for Patients Enrolled in TAILORx and RxPONDER: A Companion Protocol
Status: Not yet recruiting | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: EA1241
Record Dates: First submitted 2025-01-02; First posted 2025-01-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Submission of relapse tumor tissue specimen from biopsy confirmed cancer recurrence from patients in cohorts 1 and 2. Submission of primary tumor tissue specimen (and relapse tumor tissue if applicable from patients in cohort 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Previously enrolled on TAILORx with recurrence score (RS) 0-100 AND had a biopsy-confirmed locoregional, distant, or both locoregional and distant recurrence prior to registration on EA1241.
- Cohort 2: Previously enrolled on Step 2 of RxPONDER with recurrence score (RS) 0-25 AND had a biopsy-confirmed locoregional, distant, or both locoregional and distant recurrence prior to registration on EA1241.
- Cohort 3: Previously enrolled on Step 1 of RxPONDER and found to have a high Oncotype DX Recurrence Score (RS) 26-100.

SUMMARY:
The purpose of this study is to retrieve tissue samples from individuals with breast cancer who previously enrolled on the PACCT-1 (TAILORx) or S1007 (RxPONDER) trials and experiences a recurrence of their cancer (Cohort 1, 2, and 3), and/or the tumor initially removed at surgery in patients previously enrolled in step 1 of S1007 (RxPONDER) and found to have a high Recurrence Score of 26-100 (Cohort 3) but not followed on the study after that point. The tissue will be used for future research designed to understand why breast cancer recurs despite hormonal therapy or chemotherapy plus hormonal therapy.

DETAILED DESCRIPTION:
To collect tumor biospecimens from patients who previously enrolled in either TAILORx or RxPONDER. There are 3 separate cohorts separated by recurrence score and study:

* Cohort 1= TAILORx w/ recurrence score of 0-100
* Cohort 2= RXPONDER w/ recurrence score of 0-25
* Cohort 3= RxPONDER w/ recurrence score of 26-100

These samples will be used to assess the following primary objectives:

* Patterns of clonal evolution and the landscape of somatic alterations in paired primary tumor samples and recurrence samples
* Prevalence of the integrative cluster (IntClust) and intrinsic (PAM50) subtypes and of subtype switching in paired primary tumor samples and recurrence samples
* Identify molecular signatures, including the SET 2/3 RNA expression assay, of primary tumor specimens associated with recurrence in patients with high genomic risk and high clinical risk (Cohort 3) who received adjuvant chemotherapy plus endocrine therapy.

The study team also plans to evaluate immune composition and the prevalence of tumor-immune microenvironment (TME subtypes), and characterize the TME and cell-cell interactions in native tissue context through spatial tanscriptomic and proteomic profiling of tissue sections.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have met the criteria for 1 of the 3 possible cohorts described below:

  1. Cohort 1: Previously enrolled on TAILORx (PACCT-1) with recurrence score (RS) 0-100 AND had a biopsy-confirmed locoregional, distant, or both locoregional and distant recurrence prior to registration on this protocol.
  2. Cohort 2: Previously enrolled on Step 2 of RxPONDER (S1007) with a recurrence score (RS) of 0-25 AND had a biopsy-confirmed locoregional, distant, or both locoregional and distant recurrence prior to registration on this protocol.
  3. Cohort 3: Previously enrolled on Step 1 of RxPONDER and found to have a high Oncotype DX RS 26-100.
* Patient must have been a TAILORx (RS 0-100) or RxPONDER (RS 0-100) study participant who has the ability to understand and the willingness to sign a written informed consent document for participation in this non-intervention study (cohorts 1, 2, or 3). Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* Patient must have tumor tissue available from each cohort as outlined below:
* Patients from Cohorts 1 and 2 must have relapse tumor tissue specimen available at the time of registration for submission to ECOG-ACRIN Central Biorepository and Pathology Facility within 30 days of registration.
* Patients from Cohort 3 must have primary tumor tissue specimen available at time of EA1241 registration for submission to ECOG-ACRIN Central Biorepository and Pathology Facility within 30 days of registration

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients previously enrolled on TAILORx with a recurrence score (RS) 0-100_and RxPONDER with a recurrence score(RS) 0-25 and patients previously enrolled on RxPONDER with a recurrence score (RS) 26-100.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Patterns of clonal evolution | 2 years
  Conditional logistic regression for matched pairs, with the recurrence sample representing the case and the baseline sample the non-case in each pair, will be used to test for differences between recurrence and baseline, to estimate odds ratios, and to jointly model effects. The test for association of a single binary factor in this approach is equivalent to McNemar's test.
Prevalence of the integrative cluster (IntClust) and intrinsic (PAM50) subtypes | 2 years
  Conditional logistic regression for matched pairs, with the recurrence sample representing the case and the baseline sample the non-case in each pair, will be used to test for differences between recurrence and baseline, to estimate odds ratios, and to jointly model effects. The test for association of a single binary factor in this approach is equivalent to McNemar's test.
Molecular signatures of primary tumor specimens | 2 years
  Conditional logistic regression for matched pairs, with the recurrence sample representing the case and the baseline sample the non-case in each pair, will be used to test for differences between recurrence and baseline, to estimate odds ratios, and to jointly model effects. The test for association of a single binary factor in this approach is equivalent to McNemar's test.

SECONDARY OUTCOMES:
Immune composition | 2 years
  Evaluated using weighted Cox models
TME and cell-cell interactions | 2 years
  Evaluated using weighted Cox models
Prevalence of IntClust and PAM50 | 2 years
  Evaluated using weighted Cox models
Molecular signatures | 2 years
  Evaluated using weighted Cox models

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Sparano, MD, Principal Investigator — Eastern Cooperative Oncology Group